CLINICAL TRIAL: NCT03537339
Title: Prospective Investigation of Cardiovascular Risk Factors in Tumor Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Fei Ma, Deputy director of medical oncology, Peking Union Medical College
Other Study IDs: NCC201712029
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Cardioncology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Record general information of patients' sex, age, previous history, family history, electrocardiogram, echocardiography, cardiac biomarkers TnT, BNP, biochemical examination, and clinical treatment and so on
  Interventions: Other: Record general information

INTERVENTIONS:
Other: Record general information — Record general information of patients' sex, age, previous history, family history, electrocardiogram, echocardiography, cardiac biomarkers TnT, BNP, biochemical examination, and clinical treatment of the patients

SUMMARY:
In this study, prospective cohort study was used to collect the general information of patients' sex, age, previous history, family history, electrocardiogram, echocardiography, cardiac biomarkers TnT, BNP, biochemical examination, and clinical treatment of the patients who diagnosed cancer by pathology in National Cancer Center/ Cancer Hospital , Chinese Academy of Medical Sciences and Peking Union Medical College from January 2018 to December 2020. This study intends to evaluate and screen the cardiovascular risk of tumor patients during antitumor therapy and to establish a model of cardiovascular risk assessment for tumor patients, providing clinical evidence for the prevention of cardiovascular disease risk associated with cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of malignant tumor by pathology or cytology
2. Age 18-80, KPS > 70
3. Epidemiological information, clinical diagnosis and treatment and key information of medication are not missing.
4. The liver and kidney function were in the normal range.
5. All selected patients signed informed consent.

Exclusion Criteria:

1. patients diagnosed with congenital heart disease, cardiomyopathy, heart failure, arrhythmia, myocardial ischemia and myocardial infarction within 6 months before enrollment.
2. Severe impairment of liver and kidney function.
3. Left ventricular ejection fraction < 50% by echocardiographic examination.
4. Diagnosis of more than one kind of tumor at the same time.
5. History of surgery and trauma within 3 months before enrollment.
6. Poor compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed cancer by pathology in National Cancer Center/ Cancer Hospital , Chinese Academy of Medical Sciences and Peking Union Medical College from January 2018 to December 2020
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) related to Cardio-oncology | January 2018 to December 2020.
  Adverse events (AEs) and laboratory tests graded according to the NCI CTCAE (version 4.0) recorded by ECGs,UCGs and myocardial enzyme

CONTACTS AND LOCATIONS:
Locations (1):
- Fei Ma, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided